CLINICAL TRIAL: NCT02349113
Title: Effects of Acute Estrogen Therapy on Bone Formation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sundeep Khosla, M.D., PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 09-001935
Record Dates: First submitted 2015-01-23; First posted 2015-01-28 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Bone Loss, Age-related
Keywords: estrogen, aging
MeSH Terms: conditions — Osteoporosis | interventions — Estrogens; Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Estrogens (Experimental): Estrogens treatment: Intervention with short course (3 weeks) of treatment with transdermal estrogen (0.1mg/d)
  Interventions: Drug: Estrogens (Climara)

INTERVENTIONS:
Drug: Estrogens (Climara) — Treatment with estrogens: Estradiol dermal patch 0.1mg/d transdermally
  Other Names: Climara

SUMMARY:
This study is being done to study age-related bone changes in women. The investigators know that the major cause of osteoporosis is a shortage of the female hormone estrogen. This study will look closer at how this shortage of estrogen works to cause a decrease in bone formation.

DETAILED DESCRIPTION:
Estrogen (E) deficiency is the major cause of postmenopausal osteoporosis. Understanding the mechanisms by which E regulates bone metabolism is critical for developing novel approaches to prevent and treat this disorder. We will focus on defining mechanisms for the age-related decrease in bone formation and the role of E deficiency in mediating this decrease. We will use novel methods we have developed to examine gene expression in highly purified bone marrow osteoblastic cells. We will test whether the increase in bone formation previously observed following acute E treatment in women is associated with an increase in markers of Wnt/bone morphogenetic protein (BMP) signaling and/or production and in othe genes related to bone formation by osteoblastic cells.

ELIGIBILITY:
Inclusion Criteria:

* At least 10 years postmenopausal; Menopause is defined as no menses for at least 1 year (or documented ovariectomy) and a serum follicle-stimulating hormone (FSH) above 30 IU/L.

Exclusion Criteria:

1. Clinically significant abnormality in any of the following screening laboratory studies (to be reviewed and determined by PI or CI) : serum 25-hydroxyvitamin D (see below); phosphorus (minor change outside of normal guidelines is acceptable and does not impact the study); alkaline phosphatase and aspartate transaminase (AST) (minor change outside of normal guidelines is acceptable but not to exceed 50% above normal or ineligible); Creatinine (Cr) (minor change outside of normal guidelines is acceptable but not to exceed a value of 1.2 or ineligible); serum calcium must not exceed upper limits of normal guidelines or subject ineligible; FSH needs to be ≥30; thyroid-stimulating hormone (TSH) needs to be above 0.3 and not > 10;
2. Presence of significant liver disease, renal disease, malignancy (including breast cancer and myeloma), malabsorption syndrome, hypoparathyroidism, hyperparathyroidism, acromegaly, Cushing's syndrome, hypopituitarism, severe chronic obstructive pulmonary disease, untreated gallbladder disease, history of myocardial infarction (MI) or stroke, or history of thrombophlebitis or deep venous thrombosis;
3. Undergoing treatment with any of the following drugs: adrenocorticoid steroids (3 months or longer at anytime or > 10 days of treatment within the previous 12 months), anticonvulsant therapy (within the previous year), sodium fluoride (any history of treatment with fluoride), pharmacological doses of thyroid hormone (causing decline of TSH below normal), calcium supplementation of more than 1200 mg/d (within the preceding 3 months), bisphosphonates in the past, calcitonin (within the past six months), E therapy or treatment with a selective estrogen receptor modulator (within the past 6 months), parathyroid hormone (PTH) use in the past. Subjects with a clinical history of an osteoporotic fracture (vertebral, hip, or distal forearm) within the previous 3 years will also be excluded.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Gene expression (RNAseq analysis of gene expression from needle bone biopsies) | 3 weeks
  RNAseq analysis of gene expression from needle bone biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Sundeep Khosla, MD, Principal Investigator — Mayo Clinic

REFERENCES:
- [Derived] Farr JN, Roforth MM, Fujita K, Nicks KM, Cunningham JM, Atkinson EJ, Therneau TM, McCready LK, Peterson JM, Drake MT, Monroe DG, Khosla S. Effects of Age and Estrogen on Skeletal Gene Expression in Humans as Assessed by RNA Sequencing. PLoS One. 2015 Sep 24;10(9):e0138347. doi: 10.1371/journal.pone.0138347. eCollection 2015. PMID 26402159